CLINICAL TRIAL: NCT02015429
Title: Effect of Yellow Pea Protein and Fibre Added to a High-carb Meal on Glycemic Response and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pea_Fractionation_mixed_meal
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Diabetes
Keywords: Food intake; satiety; glycemia; appetite; blood glucose; yellow peas; fibre; protein; mixed meal
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Active Comparator): Pasta meal with added fractions or control with no fractions Pasta meal with no pea fractions
  Interventions: Dietary Supplement: Pasta meal with added fractions or control with no fractions
- 10 g protein (Experimental): Pasta meal with added fractions or control with no fractions 10 g net yellow pea protein added to pasta meal
  Interventions: Dietary Supplement: Pasta meal with added fractions or control with no fractions
- 7 g yellow pea fibre (Experimental): Pasta meal with added fractions or control with no fractions 7 g net yellow pea fibre added to pasta meal
  Interventions: Dietary Supplement: Pasta meal with added fractions or control with no fractions
- Yellow pea fibre & protein (Experimental): Pasta meal with added fractions or control with no fractions 10 g net yellow pea protein plus 7 g net yellow pea fibre added to pasta meal
  Interventions: Dietary Supplement: Pasta meal with added fractions or control with no fractions

INTERVENTIONS:
Dietary Supplement: Pasta meal with added fractions or control with no fractions

SUMMARY:
The investigators hypothesized that consuming isolated yellow pea fibre or protein, alone to together, as part of a high-carbohydrate pasta meal, would reduce the blood glucose response to the meal compared to a meal without yellow pea components and reduce food intake at a meal served 2 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* No metabolic disease
* BMI 20 - 25 kg/m^2
* male
* age 20-30

Exclusion Criteria:

* Intolerance to treatments
* on appetite-modifying medications
* restrictive eating
* smoking
* over or underweight
* breakfast-skipping

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake at second pizza meal | 135 mins after completion of treatment, 20 mins to eat pizza meal.
  Food intake measured via electronic scale in g, then converted to kcal using the caloric density.
Blood glucose | between 0 and 215 mins, every 15-30 mins
  Blood glucose measured via hand-held glucometer and finger prick.

SECONDARY OUTCOMES:
Subjective appetite | 0 to 215 minutes
  Measured via Visual Analog Scales (VAS)

OTHER OUTCOMES:
Palatability of treatments | following treatment consumption at 15 mins
  Measured by VAS to ensure palatability is not confounding other outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey G Anderson, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - University of Toronto - Department of Nutritional Sciences, Toronto, Ontario
  - University of Toronto, Toronto, Ontario